CLINICAL TRIAL: NCT06279208
Title: Exploratory Phosphoproteomic Study to Discover DYRK1A-Dependent Blood Biomarkers in TriSomy 21 Carriers
Brief Title: Phosphoproteomic Profile of Children With Down Syndrome
Acronym: PEPS
Status: Completed | Type: Observational
Sponsor: Perha Pharmaceuticals (Industry)
Collaborators: Proteas Bioanalytics (Unknown); Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A00272-43
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma from blood samples taken during a routine care consultation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Children with Down Syndrome: 30 boys with Down Syndrome, between 6 and 12 years old, coming for a routine car consultation during which blood sampling is scheduled (6 different care dedicated centers).
  Interventions: Biological: Blood sample
- Children without genetic abnormality: 30 boys without genetic abnormality, between 6 and 12 years old, coming to an analysis laboratory for a blood test (3 different laboratories)
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Recovery of plasma from the bottom of a blood collection tube.

SUMMARY:
One of the major causes of cognitive disorders limiting the learning abilities of children with Down's syndrome is excess activity of the DYRK1A protein kinase, whose gene is located on chromosome 21. Consequently, variations in the level of phosphorylation, and hence activity, of DYRK1A target proteins involved in synaptic transmission, could identify mechanisms underlying these cognitive disorders.

Several studies have shown that plasma proteins can reflect a pathophysiological brain state. The investigators plan to carry out a phosphoproteomic study to determine the phosphorylation profile of plasma proteins in children with Down's syndrome, and identify potential DYRK1A-dependent pathophysiological mechanisms and biomarkers involved in the natural course of cognition in children with Down's syndrome.

DETAILED DESCRIPTION:
During a consultation in their usual care department, dedicated to the care of children with trisomy 21, the children with trisomy 21 and their parents present will be informed about the study. An additional 2 mL of blood (from a blood sample taken as part of the consultation) will be drawn for the study by experienced nurses as part of their usual care.

Plasma from this remaining volume will be fixed and analyzed to determine a phosphoproteomic profile.

Multidimensional liquid chromatography with ultra-high resolution mass spectrometry will be used to analyze the native proteome and to obtain expression and phosphorylation levels of plasma proteins.

Similar procedure will be performed on remaining blood samples of boys without genetic abnormality having blood analysis.

Phosphoproteomic profiles of children with Down Syndrome and children without genetic abnormality will be compared to identify specific biomarkers of Down Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of free and homogeneous trisomy 21,
* Body mass index (BMI): 15-25,
* Able to understand the study based on the pictorial information leaflet and give agreement/assent to participate,
* Parent present on the day of the visit to validate their child's consent/assent, if applicable.

Exclusion Criteria:

* Celiac disease,
* Autoimmune dysthyroidism,
* Type I autoimmune diabetes,
* Alopecia,
* Other autoimmune diseases,
* Current infectious pathology,
* History of infantile spasms,
* Autism spectrum disorders,
* Epilepsy,
* Central nervous system infections,
* Leukemia not in remission,
* Anti-inflammatory treatments (NSAIDs, local or systemic corticosteroids).

Ages: 6 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: 30 Children with Down Syndrome and 30 children without genetic abnormality
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Phosphoproteomic profile | 6 months
  The main objective is to determine a phosphoproteomic signature characteristic of the pathophysiological state of trisomy 21. Plasma protein phosphorylation profiles will be analyzed using the Proteas Bioanalytics Inc. platform on blood samples taken from children with trisomy 21, and compared with the phosphorylation profiles of children without trisomy 21 of the same age and sex. Analysis and comparison of trisomy and non-trisomy phosphorylation profiles will reveal a signature characteristic of trisomy 21, potentially reflected by significant differences in plasma protein phosphorylation levels (some of which may be of cerebral origin).

SECONDARY OUTCOMES:
Identification of brain proteins | 6 months
  To determine whether the phosphoproteomic profiles characteristic of trisomy 21 make it possible to identify brain proteins (exosomes),
Impact of environnement on phosphoproteomic profile | 6 months
  To determine whether the differences potentially observed between the phosphoproteomic profiles of children with and without trisomy 21 correlate with the biological and socio-epidemiological data of children with trisomy 21,
Impact of DYRK1A on Down Syndrome specific proteomic profile | 6 months
  Determine whether the differences potentially observed between the phosphoproteomic profiles of children with and without trisomy 21 are correlated with the level of DYRK1A expression,

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - CHRU de Brest, Brest
  - CHU Grenoble, Grenoble
  - Medilab, La Châtaigneraie
  - Hospices Civils de Lyon, Lyon
  - Medilab, Niort
  - Institut Jérôme Lejeune, Paris
  - Medilab, Parthenay
  - CHU Rennes, Rennes
  - CHU Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: Undecided